CLINICAL TRIAL: NCT02247570
Title: A Randomized Controlled Trial Comparison of the Effectiveness of Carrick Brain Centers Strategies Vestibular Rehabilitation Treatment in PTSD Patients Who Have Suffered Combat Related Traumatic Brain Injuries.
Brief Title: Vestibular Rehabilitation Strategies in PTSD Effectiveness of Carrick Brain Centers Strategies Vestibular Rehabilitation Treatment in PTSD Patients Who Have Suffered Combat Related Traumatic Brain Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carrick Institute for Graduate Studies (Other)
Collaborators: Carrick Brain Centers (Industry)
Responsible Party: Principal Investigator, Frederick Carrick, PhD, FACCN, Principle Investigator, Carrick Institute for Graduate Studies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-CBC-03
Record Dates: First submitted 2014-09-18; First posted 2014-09-25 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Post Traumatic Stress Disorder PTSD
Keywords: Vestibular Rehabilitation; PTSD; DSM-IV
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vestibular Rehabilitation (Experimental): Vestibular Rehabilitation
  Interventions: Procedure: Vestibular Rehabilitation

INTERVENTIONS:
Procedure: Vestibular Rehabilitation — Stimulation of the vestibular system by off axis rotational therapy, gaze stabilization, eye movement strategies, balance training

SUMMARY:
The specific aim of this proposed study is to compare the effectiveness of Vestibular Rehabilitation (VR) in patients with PTSD who have suffered combat related traumatic brain injuries in a randomized controlled trial in terms of PTSD symptom reduction.

DETAILED DESCRIPTION:
The study has been approved by our Institutional IRB and conducted in accordance with the principles of the Declaration of Helsinki. The trial will be registered at Clinicaltrials.gov, a service of the U.S. National Institutes of Health. There is equipoise. This randomized controlled trial will compare the effectiveness of VR in in patients with PTSD who have suffered combat related traumatic brain injuries. A blinded investigator that will not be involved in the study will perform the randomization and allocation procedure.

We will accomplish the specific aim of our study by analyzing the difference in the Clinician Administered DSM-IV PTSD Scale (CAPS) scores between the two groups in our study as outcomes to compare the effectiveness of VR. The CAPS is considered to be the gold standard for diagnosing PTSD and assessing symptom severity. We expect differences in the outcomes between both treatments to be immediate and at follow-up over time, i.e. immediately after 3 months, 6 months and 12 months after cessation of a 2 week treatment period. The study design will include one pre-treatment assessment and our post-treatment assessments (at 3 months, 6 months and 12 months). Investigators who will be blinded for the allocated treatment will perform all assessments. The study will be performed at the department of Neurology of our Institutional Brain Center in Dallas, Texas. Patient recruitment will begin starting in September 2014.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with extended combat exposure, confirmed by DD-214 with combat medal and honorable discharge.
* Ages 18-60.
* Texas residents (Per funding agency).
* Medical history of TBI/head injury which occurred through military service.
* Previous medical diagnosis of PTSD or currently suffering from PTSD-like symptoms.
* Have attempted at least two of the following therapies with no significant outcome, or intolerable adverse effects: Anti-psychotic therapy (eg. Seroquel), SSRI therapy (i.e. Fluoxitiene, Celexa, etc), Atypical antidepressant therapy (Wellbutrin), Cognitive Behavior Therapy, Desensitization/exposure therapy, another form of Psychotherapy ("Talk" therapy), EMDR, or any other recognized therapy indicated for PTSD.

Exclusion Criteria:

* Concurrent therapy, including concurrent psychotherapy or pharmaceutical therapy.
* Currently addicted to alcohol or an illegal substance. If you have been through an inpatient program, you must have been released at least 90 days prior to treatment start date and have remained free from drugs and alcohol since the release from inpatient.
* Threat of harm to self and/or others
* Psychotic disorder that would prevent compliance (e.g. dissociative disorder, schizophrenia, history of catatonic states).
* Physical condition that would prevent any part of the treatment from being conducted in a safe and complete manner.
* Concussion within the last 30 days.
* History of stroke.
* Neurodegenerative disease.
* History of brain surgery, which included the removal of brain tissue.
* Previously convicted of a felony crime.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in DSM-IV CAPS | pre and post treatment and 3 months, 6 months and 1 year
  Neuropsychiatric evaluation using gold standard DSM-IV protocols

SECONDARY OUTCOMES:
Change in Computerized Dynamic Posturography | pre and post treatment and 3 months, 6 months and 1 year
  Force plate measurement of center of pressure and limits of stability
Change in Saccadometry/VNG | pre and post treatment and 3 months, 6 months and 1 year
  Measurement of visual fixation, saccades, pursuits and optokinetic responses
Change in ImPACT testing | pre and post treatment and 3 months, 6 months and 1 year
  Validated neuropsychological computerized testing

CONTACTS AND LOCATIONS:
Overall Officials: Frederick R Carrick, PhD, Principal Investigator — Carrick Brain Centers
Locations (1):
- Carrick Brain Centers, Irving, Texas, United States

IPD SHARING:
Plan to Share IPD: No